CLINICAL TRIAL: NCT06123650
Title: Post Stroke Dysphagia: Effect of Adding Brain Neuromodulation to Conventional Therapy on the Prevalence of Stroke Associated Pneumonia.
Brief Title: Post Stroke Dysphagia: Effect of Adding rTMS to Conventional Therapy on the Prevalence of Pneumonia.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Engy Badreldin Saleh Moustafa, PhD, Lecturer of Physical Therapy for Neurology and Neurosurgery, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/004748
Record Dates: First submitted 2023-11-03; First posted 2023-11-09 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2024-12

CONDITIONS: Stroke, Acute; Dysphagia; Pneumonia
Keywords: Stroke; Dysphagia; Stroke Associated Pneumonia (SAP); Repetitive Transcranial Magnetic Stimulation; Contralesional hemisphere
MeSH Terms: conditions — Stroke; Deglutition Disorders; Pneumonia

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Clinical trial, where the recruited patients will be randomly assigned into 2 equal groups ( GA & GB) using sealed envelopes, control group (GA) and study group (GB). Patients in (GA) will be treated by a designed physiotherapy program consists of: ice massage, oromotor exercises, Masako maneuver, resisted jaw opening exercise, modified chin tuck against resistance, Mandelson maneuver, effortful swallow and chin tuck in addition to sham repetitive transcranial magnetic stimulation. Patients in (GB) will be treated by low frequency (1 Hz) rTMS to the contralesional cerebral hemisphere in addition to the same Oropharyngeal physical therapy program for dysphagia as in group A.
Who Masked: Participant
Masking Description: Patients participated will be masked about the type of intervention, where (GA) patients will receive PT program + sham repetitive transcranial magnetic stimulation, while patients in (GB) will receive low frequency (1 Hz) rTMS to the contralesional cerebral hemisphere in addition to the same Oropharyngeal physical therapy program for dysphagia as in group A.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (GA) (Placebo Comparator): Group (A) will receive conventional oral care and oropharyngeal physical therapy program for dysphagia including; Exercise therapy for the oropharyngeal and tongue muscles , in addition to sham transcranial magnetic stimulation on the contralesional cerebral hemisphere.
  Interventions: Device: Sham transcranial magnetic stimulation
- Study group (GB) (Active Comparator): Group (B) will received low frequency (1 Hz) repetitive transcranial magnetic stimulation to the contralesional cerebral hemisphere in addition to the same Oropharyngeal physical therapy program for dysphagia as in group A.
  Interventions: Device: Repetitve transcranial magnetic stimulation

INTERVENTIONS:
Device: Repetitve transcranial magnetic stimulation — The Magstim Rapid2 magnetic stimulator system (Model P/N 3576-23-09, Magstim Company, Whitland, UK) was used to deliver rTMS electrical currents via a figure of 8 coil applied to the scalp against the targeted contralesional motor " Hot spot" , at a depth of approximately 1 cm . The inhibitory rTMS will be applied to the intact cerebral hemisphere at 1 Hz with a train of 1200 for 5 consecutive days.
  Arms: Study group (GB)
Device: Sham transcranial magnetic stimulation — Repetitive TMS via a sham Magstim coil (identical appearance and noise, but no active stimulation). Identical stimulation schedules as patients in study group.
  Arms: Control group (GA)

SUMMARY:
BACKGROUND: Dysphagia is one of the most life-threatening stroke complications. Dysphagic stroke patients are at increased risk of aspiration pneumonia. Pneumonia accounts for at least 10% of post stroke deaths within 30 days of hospitalization after stroke. rTMS is effective in improving post-stroke dysphagia and swallowing coordination after stimulation of the unaffected hemisphere, however it's efficacy on the prevalence of pneumonia has not yet been examined.

Purpose of the study: To determine the effect of adding low frequency repetitive transcranial magnetic stimulation to conventional oropharyngeal physical therapy program on the prevalence of aspiration pneumonia in in patients with post stroke dysphagia.

DETAILED DESCRIPTION:
Seventy acute ischemic stroke patients with oropharyngeal dysphagia from both sexes will represent the sample of this study. They will be diagnosed by a neurologist and stroke diagnosis was confirmed by brain MRI and/or CT. They will be selected from the stroke unit El Kasr El Ainy hospital, Cairo university.

Patients will be randomly assigned into two equal groups, the control group (A) and the study group (B). Control group (GA) will be treated using a designed physical therapy intervention for oropharyngeal dysphagia consists of a selected physical therapy rehabilitation program for oropharyngeal muscles in addition to sham repetitive transcranial magnetic stimulation. Study group (GB) will receive low frequency (1 Hz) rTMS to the contra-lesional cerebral hemisphere in addition to the same Oropharyngeal physical therapy program for dysphagia as in group A.

Modified Mann Assessment of Swallowing Ability (MASA) will initially used to confirm dysphagia in acute stroke. The Gugging swallowing screening (GUSS) test will be used to detect aspiration risk. A2DS2 scale will be used to detect stroke associated pneumonia (SAP). Criteria of modified Center for Disease Control and Prevention (CDC) will be used to assess SAP via assessing 4 main measures (body temperature (BT), Total Leukocyte count (TLC), Arterial blood gases (ABG), and Respiratory Rate (RR) .

The whole Intervention will consist of 12 sessions, 3 days /week for 4 consecutive weeks , Total duration of the session (TMS + PT session) will be from 40min to 60 min.

Primary & secondary outcomes will be assessed at the baseline and immediately after the completion of the whole treatment program.

ELIGIBILITY:
Inclusion Criteria:

1. All the patients were diagnosed of stroke oropharyngeal dysphagia by a neurologist. Sever to moderate dysphagia (GUSS 0-14).
2. Severity of stroke ranged from mild to moderate according to NIHSS score (NIHSS less than or equal 16).
3. Patients' age ranged from 49 to 65 years old.
4. Patients had the ability to understand and follow instructions.
5. Patients were able to sit in upright position.

Exclusion Criteria:

1. History of previous stroke.
2. History of any swallowing problem.
3. History of any head and neck surgery or tumor that causes swallowing dysfunction.
4. Any lung disease or pneumonia on admission.
5. Patients with cognitive deficits or disturbed conscious level.
6. Patients on mechanical ventilator.
7. Patients with sensory or global aphasia.

Ages: 49 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-03-22 (Actual); Primary Completion 2025-12-28 (Estimated); Study Completion 2026-01-27 (Estimated)

PRIMARY OUTCOMES:
The Gugging swallowing screen (GUSS) | Baseline and immediately after the intervention.
  It's a valid and a reliable bedside screening test to detect dysphagia and aspiration risk. The GUSS has 100% sensitivity. It begins with simple indirect swallow screen then if the total score is reached a direct swallowing test is done. It's composed of three parts: semisolid swallowing trial, liquid swallowing trial and solid swallowing trial. GUSS total score is 20. The score of the preliminary or the direct test is five. If the total score is reached the direct test can be done. Each subitem in the direct test has a score of five points. Each item of them requires the previous item to be completed.
(A2DS2) scale to detect risk of pneumonia | Baseline and immediately after the intervention.
  A2DS2 scale is used to detect stroke associated pneumonia (SAP). Consists of five items of scale which are: age, atrial fibrillation, dysphagia, sex and stroke severity. Total score of A2DS2 is 10. A2DS2 scoring tool: age more than 75 years=1, atrial fibrillation=1, dysphagia=2, male sex=1; stroke severity: is detected by NIHSS score. If NIHSS score is from 0-4=0, 5-15=3, and more than16=5. Patients with score of 6 or more are at high risk of pneumonia.
Microbiological Examination of the sputum | Baseline and immediately after the intervention
  Sputum specimens collected on sterile sputum containers by patient self-expectoration or aspiration should be checked for quality in a bacteriology laboratory. Quality check typically includes calculating the number of leukocytes (WBC) and buccal squamous epithelial (BSE) cells in the 100× view field .

SECONDARY OUTCOMES:
Body Temperature | Baseline and immediately after the intervention.
  According to the diagnostic criteria of stroke associated pneumonia (SAP):
  follow the modified Center for Disease Control and Prevention (CDC), All patients that were suspected to had pneumonia and their vitals followed the criteria of the CDC . Body temperature was one of the vitals that confirm pneumonia, Fever (>38°C) with no other recognized cause is one of the diagnostic criteria for pneumonia.
Total Leukocyte Count (TLC) | Baseline and immediately after the intervention.
  According to the diagnostic criteria of SAP follow the modified Center for Disease Control and Prevention (CDC), All patients that were suspected to had pneumonia and their vitals followed the criteria of the CDC. Leukopenia (<4000 WBC/mm3) or leukocytosis (>12 000 WBC/mm3). A blood sample is taken from the patient to assess the total leukocyte count.
Arterial Blood Gas (ABG) Test to assess Oxygen Saturation (OS) | Baseline and immediately after the intervention.
  According to the diagnostic criteria of SAP follow the modified Center for Disease Control and Prevention (CDC), All patients that were suspected to had pneumonia and their vitals followed the criteria of the CDC. TLC to assess worsening gas exchange (e.g., O2 desaturation [e.g., PaO2/FiO2≤240], increased oxygen requirements*) by taking a blood sample from the patient.
Respiratory Rate (RR) | Baseline and immediately after the intervention.
  Fast breathing was found to be the most useful sign predicting Stroke associated pneumonia (SAP) for both male and female patients .

OTHER OUTCOMES:
Mann Assessment of Swallowing Ability (MASA) | Baseline
  Screening tool for identifying eating and swallowing disorders in acute stroke , used to quantify aspiration risk via bedside test
  * predicting dysphagia and aspiration in stroke
  * 24 clinical items
  * General patient examination (alertness, cooperation, auditory comprehension, aphasia, apraxia, and dysarthria)
  * 5-point to 10-point rating scale
  * Total score: 200 points
  * cut off is 177 points
  * Risk of Dysphagia: No abnormality (≥178), mild dysphagia (168-177), moderate dysphagia (139-167), severe dysphagia (≤138)
  * Risk of Aspiration: no abnormality (≥170), mild (149-169), moderate (141-148), severe (≤140).

CONTACTS AND LOCATIONS:
Overall Officials: Engy B. Moustafa, PhD, Principal Investigator — Faculty of Physical Therapy, Cairo University, Egypt
Locations (1):
- Faculty of Physical Therapy, Cairo University, Giza, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No